CLINICAL TRIAL: NCT04667026
Title: Observational Study of Antiretroviral Therapy Cohort in Patients With HIV/AIDS
Brief Title: Observational Study on Patients With HIV/AIDS(OSPWH)
Acronym: OSPWH
Status: Recruiting | Type: Observational
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Vice chief of Infectious Disease Center, Guangzhou 8th People's Hospital
Other Study IDs: GZ8HART-v1, 20200910
Record Dates: First submitted 2020-11-19; First posted 2020-12-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; ART
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — During the study, the blood sample of patients should be preserved to detect the HIV RNA load , other co-infected microbes and drug toxicity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish a follow-up cohort of antiretroviral therapy(ART) for patients with HIV/AIDS, to observe the ART efficacy and adverse reactions, complications in the process of ART, as well as mortality and causes of death, so as to provide basis for further improving ART efficacy and quality of life of the patients.

DETAILED DESCRIPTION:
1. To establish a follow-up cohort of ART for HIV/AIDS patients: follow-up points: before treatment and 1, 2, 3 months after treatment, and every 3 months after treatment.
2. To observe the ART efficacy and adverse reactions: The clinical manifestations, laboratory and auxiliary examination indexes of each follow-up time point was observed in the follow-up cohort, including blood routine, liver function, renal function, blood lipid, blood glucose, urine routine, plasma HIV RNA,CD4 cell count, hepatitis index and syphilis index, etc. If HIV RNA is more than 1000 copies/ml, after treatment for more than 6 months, peripheral blood 10ml should be retained and drug resistance should be detected.
3. To investigate the complications of HIV/AIDS patients before and after ART.
4. To investigate the mortality and causes of death in patients with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Patients has a history of diagnosis of HIV.
* Receiving antiretroviral therapy.
* Good treatment compliance.

Exclusion Criteria:

* Aged less than 14 years of old.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HIV/AIDS who are willing to receive antiretroviral therapy.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
The rate of virological suppression after antiretroviral therapy. | Year 10
  After ART, HIV RNA level in plasma were quantified every year. The rate of HIV-RNA<400 copies/ml will be used to evaluate the efficacy of ART and the variation tendency of the rate of virological suppression will be described.

SECONDARY OUTCOMES:
The CD4+T cell counts after ART. | Year 10
  The CD4+T cell count in plasma were detected every 3 months. The variation tendency of CD4+Tcell count will be described.
All-cause mortality among HIV/AIDS after ART. | Year 10
  Describe the all-cause mortality among HIV/AIDS after ART and analyze the trend.
The incidence of adverse reactions after ART. | Year 10
  In order to assess the adverse reactions after ART, the clinical symptoms were recorded, such as respiratory symptoms, digestive system symptoms, nervous system symptoms, and mental symptoms, etc. And cytological and biochemical indexes were detected such as blood routine, liver function, renal function, blood lipid, blood glucose, urine routine, etc. Calculate the incidence of adverse reactions after ART for 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Hua Li, doctor, Principal Investigator — Guangzhou Eighth People's Hospital
Locations (1):
- Guangzhou Eighth People's Hospital, Guangzhou, Guangdong, China